CLINICAL TRIAL: NCT02126215
Title: "Blue" Cerebrovascular Reactivity (CVR) Maps as a Marker for Post-operative Delirium (POD) in Patients Undergoing Abdominal Aortic Aneurysm (AAA) Surgery: A Pilot Study: Addition of Other Patients Being Admitted to SSCU After Major Surgery
Brief Title: An MRI Study of Post-operative Delirium in Patients Undergoing Major Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Other Study IDs: B2013:057-AAA
Record Dates: First submitted 2014-04-22; First posted 2014-04-29 (Estimated); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: Postoperative Delirium
Keywords: magnetic resonance imaging; carbon dioxide; abdominal aortic aneurysm; post-op delirium
MeSH Terms: conditions — Emergence Delirium; Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study group - MRI CO2 and O2 stress test: This is a pilot study to assess feasibility of using MRI CO2 and O2 stress testing to predict POD.
  Interventions: Procedure: MRI CO2 and O2 stress testing

INTERVENTIONS:
Procedure: MRI CO2 and O2 stress testing — Pre and post operatively

SUMMARY:
Hypothesis: Patients with blue cerebrovascular reactivity (CVR) regional maps during a hypercapnic CO2 challenge will be at greater risk of developing post-operative delirium (POD) and stroke following major surgery. Blue CVR maps have also been recently documented with an O2 challenge. The blue CVR maps will be shown to be predictive of POD and stroke and ultimately represent a diagnostic test for patients at risk. These blue CVR maps will enable neurologic risk stratification for patients undergoing major surgery. Background: Major surgery is associated with a significant risk of postoperative morbidity and mortality. POD is a dreaded complication with such anesthesia and surgery. The prevalence of delirium after cardiac surgery has been reported to occur in up to 50% of patients. Using a definitive diagnostic tool such as the Confusion Assessment Method - Intensive Care Unit (CAM-ICU and CAM-S) results in the higher proportion reported. Delirium is a serious complication that results in prolonged length of stay, increased health care costs, and higher mortality. As much as $6.9 billion of Medicare hospital expenditures can be attributed to delirium. At such a cost, better diagnosis and treatment is urgently needed. Pre-emptive diagnosis leading to better management of delirium post-operatively is clearly one of the fundamental problems confronting modern anesthesia and peri-operative medicine.

Specific Objectives: The investigators seek to address (a) the identity of patients who have the greatest vulnerability to the surgery and (b) investigate the risks and test appropriate risk mitigations. Understanding POD is of immense import to help control a hospital's surgical and critical care costs. Patients with neurological consequences including POD often represent a choke point for optimized critical care utilization. At the very least, improved understanding and a diagnostic test to highlight patients at risk of POD would be most welcome. Such an advance would permit rational strategies to limit the problem and allow better designed therapeutic arcs for patients now known to be at risk. This is especially important for patients undergoing complicated major surgery and is the focus of this pilot project. Tighter control of ET respiratory gases may be indicated for both ET CO2 and ET O2 based on the results of this preliminary study.

DETAILED DESCRIPTION:
Methods: Informed witnessed consent will be obtained from all participants. Patients will have a Mini Mental State Exam (MMSE) prior to their MRI studies. A battery of neurocognitive tests will be undertaken for each subject prior to surgery. This test battery will include PHQ-9, GAD-7, Trails A and WAIS-IV Digit Span, Hopkins Verbal Learning Test Revised, Rey's Complex Figure, DKEFS, F-A-S, CLOX I and II. This will take 45-60 minutes. Patients will have CVR maps with blood oxygen level dependent (BOLD-MRI) pulse sequences done with standard RespirAct (a computer-controlled gas blender) protocols in association with anatomic imaging in a 3.0 Tesla magnet. The clinical care team and patient will be blinded as to the CVR results. Patients will have standardized anesthesia and per usual approaches for their major surgery and have standard POD assessment tools (CAM-ICU and CAM-S). Storage of anesthesia hemodynamics will be to digital data acquisition systems for later collation. End-tidal CO2 will be targeted at patient baseline values +/- 2.5 mmHg during the surgical procedure and if ventilated for any period post-operatively. Inspired O2 will be targeted to 0.3 - 0.6, based on pulse oximetry of greater than 95% with adequate arterial oxygenation confirmed by ABG. Standard fast-track protocols and admission to the surgical special care unit (SSCU) will be undertaken to facilitate patient management. Any patient with obvious POD, post-op delirium or stroke will be managed per usual protocols. Multiple CVR maps (650 studies) have been done at University Health Network in Toronto. As well over 150 studies have been conducted at the Health Sciences Centre at the University of Manitoba in the past 5 years.

Significance/Importance: This study has the potential to make an important contribution in the understanding of POD for all surgical procedures and specifically a window into the problem with major surgery. A positive study based on our hypothesis can fundamentally change our understanding of cognitive dysfunction after surgery. Large follow-up multicentre trials can be constructed based on initial findings from this pilot study if the study bears fruit. At the least, further elucidation into POD for major surgery is expected with this study. tighter control of end-tidal gases may be a consequence of the findings of this study.

ELIGIBILITY:
Inclusion Criteria:

* major surgery
* able to tolerate CO2 and O2 stress test

Exclusion Criteria:

* diagnosed dementia
* unable to have MRI
* excessive claustrophobia
* unstable angina, recent myocardial infarction (MI)
* chronic obstructive pulmonary disease (COPD)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled to undergo major surgery.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2014-07; Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Blue voxel count/whole brain voxel count | Baseline
  the number and distribution of 'blue' voxels - those with reversed CO2 and O2 responsiveness to a controlled CO2 and O2 change with blood oxygen level dependent (BOLD) MRI.
Incidence of post-op delirium | Post-op out to discharge or maximum of 2 weeks post-surgery
  the incidence and severity of post-op delirium using the cognitive assessment method - intensive care unit (CAM-ICU) scoring approach twice a day.

SECONDARY OUTCOMES:
Length of Stay (LOS) in hospital | post-operatively to 2 weeks
  Length of stay in hospital - number of days from day of surgery up to a maximum of 2 weeks.
Stroke | Post-op until time of discharge up to 2 weeks
  Post-op stroke rate and severity will be assessed.
Intra-operative blood pressure | Intra-operative
  Blood pressure will be measured in mmHg at 60 hz. during the operative procedure. The nadir and time below 60 mmHg will be recorded.

OTHER OUTCOMES:
Pre-op test for post-operative delirium (POD) | up to 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: W. Alan Mutch, MD, Principal Investigator — University of Manitoba
Locations (1):
- Kleysen Institute for Advanced Medicine - Health Sciences Centre, Winnipeg, Manitoba, Canada

REFERENCES:
- [Background] Mutch WA, Mandell DM, Fisher JA, Mikulis DJ, Crawley AP, Pucci O, Duffin J. Approaches to brain stress testing: BOLD magnetic resonance imaging with computer-controlled delivery of carbon dioxide. PLoS One. 2012;7(11):e47443. doi: 10.1371/journal.pone.0047443. Epub 2012 Nov 5. PMID 23139743
- [Background] Mutch WAC, El-Gabalawy R. Anesthesia and postoperative delirium: the agent is a strawman - the problem is CO2. Can J Anaesth. 2017 Jun;64(6):678-680. doi: 10.1007/s12630-017-0859-3. Epub 2017 Mar 10. No abstract available. PMID 28283991
- [Background] El-Gabalawy R, Patel R, Kilborn K, Blaney C, Hoban C, Ryner L, Funk D, Legaspi R, Fisher JA, Duffin J, Mikulis DJ, Mutch WAC. A Novel Stress-Diathesis Model to Predict Risk of Post-operative Delirium: Implications for Intra-operative Management. Front Aging Neurosci. 2017 Aug 18;9:274. doi: 10.3389/fnagi.2017.00274. eCollection 2017. PMID 28868035
- [Background] Mutch WAC, El-Gabalawy RM, Graham MR. Postoperative Delirium, Learning, and Anesthetic Neurotoxicity: Some Perspectives and Directions. Front Neurol. 2018 Mar 20;9:177. doi: 10.3389/fneur.2018.00177. eCollection 2018. PMID 29615969
- [Background] Mutch WAC, El-Gabalawy R, Girling L, Kilborn K, Jacobsohn E. End-Tidal Hypocapnia Under Anesthesia Predicts Postoperative Delirium. Front Neurol. 2018 Aug 17;9:678. doi: 10.3389/fneur.2018.00678. eCollection 2018. PMID 30174647
- [Derived] Mutch WAC, El-Gabalawy R, Ryner L, Puig J, Essig M, Kilborn K, Fidler K, Graham MR. Brain BOLD MRI O2 and CO2 stress testing: implications for perioperative neurocognitive disorder following surgery. Crit Care. 2020 Mar 4;24(1):76. doi: 10.1186/s13054-020-2800-3. PMID 32131878